CLINICAL TRIAL: NCT03634306
Title: A Randomized, Controlled Study Evaluating The Effectiveness Of The Ultravision Visual Field Clearing System in Laparoscopic Hysterectomy and Myomectomy
Brief Title: Ultravision Visual Clearing System in Laparoscopic Hysterectomy and Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, David Levine, Director Minimally Invasive Gynecology, Mercy Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18-091
Record Dates: First submitted 2018-06-28; First posted 2018-08-16 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-01

CONDITIONS: Pain; Hysterectomy; Myomectomy
Keywords: Visual clearing System Laparoscopic Hysterectomy Myomectomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: STUDY DESIGN This is a prospective blinded, randomized controlled study. Arms 1 and 2: Patients enrolling in study arms 1 and 2 who are undergoing hysterectomy will be randomized to either the Ultravision™ System (Arm 1) or Standard of Care/no Ultravision (Arm 2) study arms.
  Arm 3: Patients enrolling in study arm 3 who are undergoing a myomectomy will have their procedure conducted with the Ultravision™ System. The procedure is purported to generate the greatest smoke and therefore constitutes a worst-case challenge for the system.
  All prescribed evaluations will be performed for all study arms.
  STUDY SIZE Arms 1 and 2 (randomized) will enroll 15 patients each. Arm 3 will enroll an additional 5 patients.
  DURATION The total duration of the study is expected to be approximately 6 months.
Who Masked: Investigator
Masking Description: Patients will be randomized using a paper envelope system, just prior to surgery. Investigator will not be informed of the randomization assignment until after the patient is discharged (end of follow-up period). A simple envelope system is used. Pre-made study arm assignment envelopes will be created. Envelopes will be opened just prior to the procedure. For patients randomized & withdrawn prior to the procedure or converted to open procedure, replacement envelopes will be added to the envelope pool. To preserve blinding during the procedure, the Ultravision System consumable will be introduced into the patient, generator will appear operational during all procedures. The display will be covered during use so the investigator is not aware the system is on/off. If for any reason un blinding occurs, the reason will be recorded. Study assessments will be collected per protocol, but the data will not be pooled with blinded data for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- ARM 1 (Active Comparator): Laparoscopic hysterectomy with use of the Ultravision System
  Interventions: Device: Ultravision System
- ARM 2 (Placebo Comparator): Laparoscopic Hysterectomy per Standard of Care/no Ultravision System
  Interventions: Procedure: Laparoscopic Hysterectomy
- ARM 3 (Active Comparator): Laparoscopic myomectomy with use of the Ultravision System.
  Interventions: Device: Ultravision System

INTERVENTIONS:
Device: Ultravision System — Laparoscopic surgery will be performed with the Ultravision Visual Field Clearing System. This system is indicated for the clearance of smoke and other particulate matter that is created during laparoscopic surgery. Ultravision Visual Clearing System removes surgical smoke by means of electrostatic precipitation.
  Arms: ARM 1; ARM 3
Procedure: Laparoscopic Hysterectomy — Laparoscopic hysterectomy will be performed according to standard of care without the Ultravision Visual Field Clearing System
  Arms: ARM 2

SUMMARY:
This is a prospective blinded, randomized controlled study. The study will include three study arms:

Patients undergoing laparoscopic hysterectomies will be randomized to one of either "Ultravision" (study arm 1) or "no Ultravision" (study arm 2, i.e. the current standard of care) groups. The study will be conducted blinded to the investigator during the procedure through patient discharge. The Ultravision system will be present in both, with the generator covered (not seen by user) and either on or off depending on the randomization. 30 patients will be enrolled, 15 per group. Five patients undergoing myomectomy will have their procedures conducted using the Ultravision (study Arm 3).

Ultravision is cleared for use in all laparoscopic surgery i.e. including laparoscopic hysterectomy and myomectomy, in the United States. However, the clinical benefits arising from its use in gynecology have not yet been quantitatively assessed and published in an independent medical journal.

Study Purpose:

There are three main study objectives

1. To evaluate the impact of use of Ultravision device during laparoscopic hysterectomy and myomectomy on the quality of visualization in the laparoscopic field
2. To evaluate the impact of use of Ultravision device during laparoscopic hysterectomy and myomectomy on procedural characteristics
3. To evaluate the impact of use of Ultravision device during laparoscopic hysterectomy and myomectomy on clinical outcomes.

DETAILED DESCRIPTION:
Background: The smoke generated by electrosurgical devices in the process of dissection of tissues during laparoscopy can obscure the surgical visual field. Laparoscopic hysterectomy and laparoscopic myomectomy are procedures that produce a considerable amount of smoke, which impedes the operating surgeon. It is often necessary to suspend the surgery to allow the smoke to dissipate, or more commonly open a laparoscopic port to vent the smoke into the room, adding to the operating time. It is also common to remove the laparoscope to clean the lens because it can be soiled by the smoke as well. In order to enhance the dissipation of smoke and maintain an adequate pneumoperitoneum it is often necessary to increase the flow of carbon dioxide (CO2) from the insufflator. Surgical smoke handling during laparoscopic surgery results in an increase of the known risks to the patient of using excessive CO2; as well exposing the operating room staff to the smoke which may create a potential health concern. The electrostatic-precipitation of laparoscopic smoke is a new technique, marketed under the name Ultravision©, making it possible to precipitate the smoke as it is created, thereby actively eliminating it from the field of view. Safety and feasibility studies have been carried out allowing it to be placed on the market in Europe, Japan and the United States. A randomized study of its clinical effectiveness (ref: Ansell J. Surg, Endosc. (2014) 28: 2057-2065) showed that electrostatic-precipitation significantly improved visibility (reduction of visual impairment) and reduced surgery time in laparoscopic cholecystectomy. Ultravision is cleared for use in all laparoscopic surgery i.e. including laparoscopic hysterectomy and myomectomy, in the United States. However, the clinical benefits arising from its use in gynecology have not yet been quantitatively assessed and published in an independent medical journal.

Study Purpose: here are three main study objectives;

1. To evaluate the impact of use of Ultravision device during laparoscopic hysterectomy and myomectomy on the quality of visualization in the laparoscopic field
2. To evaluate the impact of use of Ultravision device during laparoscopic hysterectomy and myomectomy on procedural characteristics
3. To evaluate the impact of use of Ultravision device during laparoscopic hysterectomy and myomectomy on clinical outcomes.

Primary Hypothesis: The primary hypothesis being tested in this study is that using Ultravision during laparoscopic hysterectomy and myomectomy improves visualization similar to that reported when used in laparoscopic cholecystectomy without the need for CO2 exchange and that, by doing so, the amount of CO2 that the patient is exposed to is reduced compared to the current standard of care.

Secondary hypothesis: There are two aspects to CO2 exposure during laparoscopic surgery: the amount of gas used and the intra-abdominal pressure of the pneumoperitoneum. Ultravision has already been shown in laparoscopic cholecystectomy to minimize the amount of CO2 that a patient is exposed to during laparoscopic surgery because it does not rely on the process of dilution using ongoing CO2 supply from the insufflator. Decreasing the intra-abdominal pressure below the conventional 12-15 mmHg during laparoscopic surgery has been shown by others to lead to improved clinical outcomes in other laparoscopic procedures.

In this study the target abdominal pressure for all procedures conducted will be 10mmHg. The ability to maintain that pressure during the procedure in the different study arms will be reported and compared. In addition to this secondary endpoint other procedure data will be collected to assess the potential impact of the Ultravision technology on procedure characteristics such as adverse events, procedure time, patient temperature, patient end tidal CO2 level, post-op medications for pain etc.

INTENDED USE: The Ultravision™ System is indicated for the clearance of smoke and other particulate matter that is created during laparoscopic surgery.

DEVICE DESCRIPTION: The Ultravision™ System is an accessory to electrosurgical instruments that is used to clear the surgical smoke generated during their use and as such will only be used when such devices are in use. An example of the effect of the Ultravision™ System during use to improve the visualization of the field of view.

The system includes the following elements: Standalone battery-operated generator unit Ionwand™, which is introduced into the abdomen of the patient through either the Ultravision™ 5mm Trocar or a 2.5mm percutaneous catheter and provides the source of the electrons that create the negative ions that transiently charge the surgical smoke particles. Other accessories include a patient return adaptor and battery recharging station.

US REGULATORY STATUS: The Ultravision™ System obtained regulatory clearance through US FDA's De Novo Classification Process (DEN 150022). The system has been in distribution in Europe since January 2014 and in the US since December of 2016, over 250 systems are currently in use. To date there have been no incident or medical device reports (patient injury reports) and there have been no product recalls.

SUBJECT IDENTIFICATION & SELECTION: Potential subjects will be identified from the clinical practice of the participating investigator or by their respective research staff. Each new subject presenting for evaluation or inclusion is to be assessed for adherence to the following inclusion/exclusion criteria. Patients are considered enrolled once it has been demonstrated that the inclusion/exclusion criteria have been met and the patient signs the informed consent.

SUBJECT INFORMED CONSENT: Referred patients presenting for diagnosis or treatment consistent with the inclusion criteria will undergo the informed consent process.

PREOPERATIVE PROTOCOL: Patients will be assessed preoperatively in accordance with the current standard of care. The Ultravision™ System will be set up in the OR for all cases. For randomized study arms 1 and 2, the system will be covered such that the electronic display is not visible to the investigator. The system will be turned off for all non-Ultravision procedures. For all procedures, the Ionwand will be inserted/introduced as described in the Instructions for Use.

SURGEON VISUALIZATION SURVEY: Immediately post procedure the investigator will be asked three questions:

1. Proportion of operating time with effective visibility? A 1-100 visual analog scale will be used to estimate the time proportion.
2. What is the overall rating of visibility?
3. For randomized study arms do you know if the patient was in the Ultravision group? A yes or no, or don't know answer and the information that influenced the answer is recorded.

POST PROCEDURE FOLLOW-UP PROTOCOL: Post procedure follow-up assessments include discharge and 2-week follow-up, which is the current standard of care.

ADVERSE EVENT CATEGORIES: For purposes of this protocol the adverse event definitions are derived from Good Clinical Practice (GCP) standards and FDA Guidance.

The signs, symptoms, and sequelae of an underlying adverse event (linked pathophysiologically to the AE) should not be reported as separate adverse events. All adverse events, of any type, are to be recorded on an "Adverse Event Form". Adverse events are to be characterized by their severity, relatedness the implant procedure, need for therapy, and resolution status.

Adverse events will initially be characterized as "serious" or "non-serious" by the study investigator.

ADVERSE EVENT ADJUDICATION: Events are to be initially judged by the investigator as to their relatedness to the study device, implant procedure, or "other etiology". The classifications will be "not related", "probably not related", "undetermined", "probably related", or "related".

REPORTING OF ADVERSE EVENTS AND UNANTICIPATED PROBLEMS Serious adverse events and Unanticipated Problems related to the research will be reported to the Mercy Institutional Review Board.

SUBSEQUENT SURGICAL INTERVENTIONS: Some complications may lead to a subsequent surgical intervention. The reason for each subsequent surgical intervention and the action taken is recorded on the case report form, along with the identification of the type subsequent surgical interventions according. The exact type of intervention must be specified.

PATIENT WITHDRAWAL: A patient may choose to withdraw from participation in the study at any time without penalty. If a patient chooses to withdraw they will still receive medical care consistent with the standard of care. The investigator may at their discretion withdraw a patient from participation. Examples include if the procedure necessitates conversion from laparoscopic to open technique, lack of adherence to visit schedule, adverse events, or safety concerns. For all withdrawals the date, point in the study, and reason for withdrawal will be recorded.

STUDY SUSPENSION/TERMINATION: If for any reason the principle investigator chooses to suspend or terminate the study, the IRB shall be informed of the decision and the basis of the decision.

PROVISION AND INVENTORY OF STUDY DEVICES: The device and required materials will be provided to the Investigator by Alesi Surgical Ltd.

DATA COLLECTION AND MANAGEMENT: The investigators are responsible for collecting the data from the study.

IMAGING DIAGNOSTICS: All imaging performed for patients is considered consistent with standard of care.

SAMPLE SIZE JUSTIFICATION: The sample size selected (15) per group is considered to be a number to allow for a meaningful comparison between the study arms conducted by a single investigator. As a post-market study intended to evaluate user satisfaction and relative impact the Ultravision™ System has on the procedure as opposed to demonstrating safety and efficacy, the sample size is considered to be sufficient for that purpose. This essential information is identified in the primary and secondary endpoints.

DATA ANALYSIS; Data collected will be summarized using descriptive statistics. For study success results must demonstrate a clinical benefit for the randomized Ultravision group compared to the no Ultravision group based upon the primary endpoint analysis. Additional exploratory analysis may be conducted during data analysis. Because the study is not statistically powered, analysis for primary and secondary endpoints will be conducted using comparative statistics with the caveat understood regarding the relatively small sample sizes for each group.

ADMINISTRATION: This study is being conducted as an "Investigator Sponsored" post-market study. The Investigator holds ultimate responsibility for the design, conduct, analysis, and reporting of the results from this study and is the primary contact for all matters related to this investigational plan. The Primary Investigator is also accountable for monitoring this investigation and performing those actions necessary to protect the scientific credibility of the way this study is conducted.

REGULATORY COMPLIANCE: The investigators and all research staff participating in this investigation are expected to adhere to this investigational plan, Good Clinical Practices, applicable privacy laws, the Declaration of Helsinki, and any approval requirements imposed by an Institutional Review Board. The study will be submitted for review and approval by the Mercy Institutional Review Board.

PRIVACY AND CONFIDENTIALITY: This study is to be performed in accordance with all applicable privacy laws. All data and information concerning subjects and their participation in this trial are considered confidential. Only authorized investigators and approved study personnel will have access to some portions of these confidential files. Institutional Review Boards and other regulatory authorities also have the right to inspect and copy records pertinent to this trial. All public reporting of the results of this study will eliminate identifiable references to the subjects.

RISK/BENEFIT ASSESSMENT: As a surgical accessory device, the Ultravision™ System does not administer any medical treatment. The risks associated with its use are consistent with other surgical accessories used in laparoscopic surgery. The device has been tested for sterility, biocompatibility, and electrical safety demonstrating that such risks have been mitigated to acceptable levels.The benefits that are being evaluated in this study are improved visualization, lower pressure of pneumoperitoneum, and CO2 consumption have the potential to favorably impact patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST meet all the following:

* Is 21 years or older.
* Provide written informed consent prior to trial procedures after studies indicate that the patient needs the prescribed procedure.
* Agrees to attend all follow-up assessments.
* Is clinically indicated to undergo laparoscopic hysterectomy or myomectomy.

Exclusion Criteria:

* Subjects MUST not have any of the following:

  * Existing comorbidities that would contraindicate them for laparoscopic surgery.
  * Be pregnant.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will enroll female patients who are indicated for laparoscopic hysterectomy or myomectomy.
Enrollment: 35 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Levine, MD, Principal Investigator — Mercy Research
Locations (1):
- Mercy Hospital St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARM 1 | ARM 2 | ARM 3
Started | 15 | 15 | 5
Completed | 15 | 15 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 1 | ARM 2 | ARM 3 | Total
Number analyzed (Participants) | 15 | 15 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.2) | 46.1 (8.5) | 37.2 (9.7) | 44.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 5 | 35
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 11 | 12 | 2 | 25
  Black/African-American | 4 | 2 | 3 | 9
  Hispanic/Latino | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 5 | 35
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 30.4 (7.2) | 33.3 (10.5) | 32.7 (9.7) | 32.0 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Surgical Field Visualization
Description: Measure the quality of visualization in the laparoscopic field of view using a 5 point Visual Analog Scale. 0 is visible interference is imperceptible, 2-3 is perceptible to interfering, 4 is interfering, 5 is highly interfering)
Time Frame: End of procedure
Measure: Number; unit: participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
participants
  Imperceptible Visual Impairment | 9 | 1 | 5
  Perceptible Visual Impairment | 2 | 2 | 0
  Slightly Interfering | 3 | 7 | 0
  Interfering | 1 | 4 | 0
  Highly Interfering | 0 | 1 | 0

2. Primary Outcome: Consumed CO2
Description: Amount of CO2 Consumed in liters from placement of all surgical ports to colpotomy (hysterectomy) or closure of last uterine defect (myomectomy)
Time Frame: End of procedure
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Liters | 16.7 (21.3) | 23.5 (23.7) | 25.7 (25.3)

3. Secondary Outcome: Operative Procedure Disruption
Description: Count of the number of times the operative procedure is interrupted or delayed due to clearing smoke
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Count of pauses for smoke clearing
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Count of pauses for smoke clearing | 1.6 (1.7) | 3.6 (2.2) | 0 (0)

4. Secondary Outcome: Intra-abdominal Pressure
Description: Maximum intra-abdominal pressure used measured in mmHg
Time Frame: End of procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
mmHg | 10.7 (1.8) | 12.3 (2.6) | 10 (0)

5. Secondary Outcome: Number of Participants With Adjusted Intra-abdominal Pressure
Description: The number of participants who had an adjustment in intra-abdominal pressure during the procedure
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 2 | 7 | 0

6. Secondary Outcome: Duration of Intra-abdominal Pressure Increase
Description: Duration spent at first intra-abdominal pressure increase from the initial 10mmHg set point
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
minutes | 31.5 (6.4) | 59.8 (37.4) | 0 (0)

7. Secondary Outcome: Temperature at Time 0 Min
Description: Temperature in degrees Celsius at time 0 min during operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Degrees Celsius | 35.93 (0.49) | 35.75 (0.51) | 35.96 (0.48)

8. Secondary Outcome: Temperature at Time 15 Min
Description: Temperature in degrees Celsius at 15 min during operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Degrees Celsius | 35.93 (0.44) | 35.87 (0.30) | 36.14 (0.39)

9. Secondary Outcome: Temperature at Time 30 Min
Description: Temperature in degrees Celsius at 30 min during operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Degrees Celsius | 35.99 (0.48) | 35.93 (0.29) | 36.18 (0.33)

10. Secondary Outcome: Temperature at Time 45 Min
Description: Temperature in degrees Celsius at 45 min during operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Degrees Celsius | 36.03 (0.51) | 36.09 (0.36) | 36.42 (0.22)

11. Secondary Outcome: Temperature at Time 60 Min
Description: Temperature in degrees Celsius at 60 min during operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 14 | 15 | 5
Degrees Celsius | 36.19 (0.52) | 36.05 (0.30) | 36.20 (0.40)

12. Secondary Outcome: End-Tidal CO2 Level at Time 0
Description: End-Tidal CO2 leve; recorded at 0 min during the operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Percent CO2
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Percent CO2 | 35.4 (3.0) | 35.1 (2.6) | 33.6 (2.0)

13. Secondary Outcome: End-Tidal CO2 Level at Time 15
Description: End-Tidal CO2 level recorded at 15 min during the operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Percent CO2
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Percent CO2 | 35.7 (3.7) | 36.1 (2.4) | 34.2 (1.3)

14. Secondary Outcome: End-Tidal CO2 Level at Time 30
Description: End-Tidal CO2 level recorded at 30 min during the operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Percent CO2
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Percent CO2 | 35.1 (4.2) | 35.8 (3.4) | 34.0 (1.0)

15. Secondary Outcome: End-Tidal CO2 Level at Time 45
Description: End-Tidal CO2 level recorded at 45 min during the operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Percent CO2
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Percent CO2 | 35.9 (2.8) | 35.4 (3.5) | 35.4 (1.7)

16. Secondary Outcome: End-Tidal CO2 Level at Time 60
Description: End-Tidal CO2 level recorded at 60 min during the operative procedure
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Percent CO2
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 14 | 15 | 5
Percent CO2 | 36.1 (3.1) | 35.0 (2.8) | 35.8 (1.6)

17. Secondary Outcome: Duration of Procedure
Description: Time from placement of last surgical port to colpotomy (hysterectomy) or closure of last uterine defect (myomectomy)
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Minutes | 40.5 (20.8) | 46.9 (18.3) | 56.8 (31.5)

18. Secondary Outcome: Number of Participants With a Hospital Stay Less Than 24 Hours
Description: The number of participants with a hospital duration of stay less than 24 hours recorded as "yes" or "no." Data represent the number of participants with a hospital stay less than 24 hours.
Time Frame: 2 weeks following procedure completion
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 15 | 15 | 5

19. Secondary Outcome: Postoperative Pain Numerical Rating Scale
Description: Post operative pain evaluated according to a numerical rating scale from 0 (no pain) to 10 (worst pain possible)
Time Frame: Before hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
score on a scale | 2.7 (2.4) | 2.7 (1.8) | 2.8 (1.9)

20. Secondary Outcome: Postoperative Pain Numerical Rating Scale
Description: Post operative pain evaluated according to a numerical rating scale from 0 (no pain) to 10 (worst pain possible)
Time Frame: 2 weeks following procedure completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
score on a scale | 0.7 (2.3) | 0.1 (0.5) | 0 (0)

21. Secondary Outcome: Number of Participants That Received Post-operative Opioid Pain Medication
Description: The number of participants that received post-operative opioid pain medication during hospital stay recorded as "yes" or "no." Data represent the number of participants that received post-operative opioid pain medication during hospital stay.
Time Frame: Post-operative hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 12 | 12 | 5

22. Secondary Outcome: Number of Participants That Received Post-operative Non-opioid Pain Medication
Description: The number of participants that received post-operative non-opioid pain medication during hospital stay recorded as "yes" or "no." Data represent the number of participants that received post-operative non-opioid pain medication during hospital stay.
Time Frame: Post-operative hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 14 | 14 | 5

23. Secondary Outcome: Number of Participants Reporting Opioid Pain Medication Use at Follow up
Description: The number of participants that reported opioid pain medication use at follow up visit recorded as "yes" or "no." Data represent the number of participants that reported opioid pain medication use at follow up.
Time Frame: 2 week follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 10 | 7 | 5

24. Secondary Outcome: Number of Participants Reporting Non-opioid Pain Medication Use at Follow up
Description: The number of participants that reported non-opioid pain medication use at follow up visit recorded as "yes" or "no." Data represent the number of participants that reported non-opioid pain medication use at follow up.
Time Frame: 2 week follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 10 | 9 | 1

25. Secondary Outcome: Adverse Events Related to Procedure
Description: Number of subjects with adverse events determined probably related or related to procedure
Time Frame: Intraoperative up to 2 weeks post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 5 | 2 | 0

26. Secondary Outcome: Adverse Events Related to Smoke Clearing Device
Description: Number of subjects with adverse events determined probably related or related to smoke clearing device
Time Frame: Intraoperative up to 2 week follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 | ARM 2 | ARM 3
Number analyzed (Participants) | 15 | 15 | 5
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from screening/baseline through the 2-week follow up visit.
Arm/Group | ARM 1 | ARM 2 | ARM 3
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 5/15 | 9/15 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 (N=15) | ARM 2 (N=15) | ARM 3 (N=5)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) — Inability to urinate
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Elevated platelet count
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Mood changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bell's Palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Concomitant planned breast surgery
Bladder Perforation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) — Intra-operative identification and removal of ovarian mass
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Intra-operative identification and removal of cyst
Endometriosis lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Intra-operative identification and removal of endometriosis lesion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03634306/Prot_SAP_000.pdf